CLINICAL TRIAL: NCT06770192
Title: Effects of Plyometrics and Calisthenics on Executive Function in School Going Children
Brief Title: Comparison Between Plyometrics and Calisthenics on Executive Function in School Going Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RiphahRCRAHS-ISBRECMS-PT01917
Record Dates: First submitted 2024-12-12; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Executive Function
Keywords: Executive function; Calisthenics; Plyometric exercises; School-going children; Cognitive development; Physical activity; Working memory; Selective attention; Inhibitory control; Cognitive flexibility; Stroop test; Trail Making Test; Digit Span Test; Cognitive assessment in children
MeSH Terms: conditions — Motor Activity | interventions — Gymnastics; Plyometric Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Plyometric (Experimental): Session will start with 9 minutes of warm up which includes 4 minutes of jogging and moderate intensity dynamic stretching for 5 minutes.. And 9 minutes cool down period. Following Plyometrics would be performed:1 medicine ball squats 2.ABC pushups 3.Medicine ball chest press 4.standing jump reach for star 5.SINGLE leg hops 6.Pushup on knees 7.zig zag double jump
  Interventions: Other: Plyometric
- Calisthenics (Experimental): Session will start with 9 minutes of warm up which includes 4 minutes of jogging and moderate intensity dynamic stretching for 5 minutes. Session would be of 8 minutes in which 1 minutes exercise and 1 minute rest is there. Exercise include bunny jumps, bear crawls , crab walk and mad cat and 9 minutes cool down period. This protocol would be follow up to 8 weeks.
  Interventions: Other: Calisthenics
- Control (Other): compare with other groups
  Interventions: Other: Control

INTERVENTIONS:
Other: Calisthenics — Session will start with 9 minutes of warm up which includes 4 minutes of jogging and moderate intensity dynamic stretching for 5 minutes. Session would be of 8 minutes in which 1 minutes exercise and 1 minute rest is there. Exercise include bunny jumps, bear crawls , crab walk and mad cat and 9 minutes cool down period. This protocol would be follow up to 8 weeks.
  Arms: Calisthenics
Other: Plyometric — : Session will start with 9 minutes of warm up which includes 4 minutes of jogging and moderate intensity dynamic stretching for 5 minutes.. And 9 minutes cool down period. Following Plyometrics would be performed:1 medicine ball squats 2.ABC pushups 3.Medicine ball chest press 4.standing jump reach for star 5.SINGLE leg hops 6.Pushup on knees 7.zig zag double jump
  Arms: Plyometric
Other: Control — compare with other groups
  Arms: Control

SUMMARY:
The goal of this clinical trial is to compare the effects of calisthenics and plyometric exercises on executive functions in school-going children. The main questions it aims to answer are:

* Will calisthenics exercises have a better effect on executive functions compared to plyometric exercises in school-going children?
* How do these exercise interventions impact selective attention, working memory, inhibitory control, and cognitive flexibility in children?

Researchers will compare a calisthenics exercise group, a plyometric exercise group, and a control group (no intervention) to see if there are differences in executive function outcomes.

Participants will:

* Be male school-going children aged 8-12 years
* Be randomly assigned to one of three groups: calisthenics, plyometric, or control
* Complete baseline assessments of executive function
* Participate in their assigned exercise program 3 times per week for 8 weeks (exercise groups only)
* Complete follow-up assessments of executive function at 4 weeks and 8 weeks
* Perform tests measuring selective attention, working memory, inhibitory control, and cognitive flexibility

DETAILED DESCRIPTION:
Title: Comparison of Calisthenics and Plyometric Exercises on Executive Functions Among School-Going Children

This research study, conducted by Maria Javid at Riphah International University in Islamabad, aims to investigate how different types of exercise affect cognitive abilities in children. Specifically, it compares the effects of calisthenics (bodyweight exercises) and plyometrics (jump training) on executive functions in school-going children.

Executive functions are crucial cognitive skills that help children with tasks like planning, organizing, paying attention, and controlling impulses. These skills are essential for academic success and everyday life. The study seeks to understand if and how different exercise types can enhance these cognitive abilities.

Key Details:

* Participants: Male school-going children aged 8-12 years
* Duration: 8 weeks
* Location: Public and private schools in Islamabad, Pakistan

The study will involve three groups:

1. Calisthenics group: Performing bodyweight exercises
2. Plyometric group: Engaging in jumping and explosive movement exercises
3. Control group: No specific exercise intervention

Both exercise groups will participate in supervised sessions three times per week. The exercises are designed to be age-appropriate and safe for children.

Measurements:

Researchers will assess various aspects of executive function using standardized tests:

* Selective attention: Using the Children's Trail Making Test
* Working memory: Using Forward and Backward Digit Span Tests
* Inhibitory control and cognitive flexibility: Using the Stroop Test

These assessments will be conducted at the beginning of the study, at 4 weeks, and at 8 weeks to track changes over time.

Significance:

This study is important because it could provide valuable insights into how different types of exercise affect children's cognitive development. The results could inform physical education programs in schools and help parents and educators make informed decisions about children's physical activities.

Ethical Considerations:

The study has been approved by the university's ethics review board. Participation is voluntary, and parents must provide informed consent. All data will be kept confidential and coded to protect participants' identities.

Expected Outcomes:

The researchers hypothesize that calisthenics exercises may have a more significant positive effect on executive functions compared to plyometric exercises. However, both exercise types are expected to show improvements compared to the control group.

This research contributes to the growing field of exercise neuroscience and could have practical implications for child development, education, and public health policies related to physical activity in schools.

ELIGIBILITY:
Inclusion Criteria:

* Participants falling in this category would be recruited into the study.
* Male School Going Children (8-12 Years of Age)
* Normal BMI of School Going Children
* No Recent Musculoskeletal Injury.
* Not Actively Engaged in Other Sports

Exclusion Criteria:

* Children with any mental or physical disability.
* Children with acute illness or fracture
* Active Inflammation or infections
* Any physical deformity

Ages: 8 Years to 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — male participants are eligible to enroll in the study
Enrollment: 99 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-04-04 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
Selective Attention | 8 weeks
  which is measured by Children's Trail Making Test (Parts 1 and 2).Part 1: This test assesses the child's ability to maintain focused attention by having them connect numbered circles in sequential order as quickly as possible. It measures visual attention and task-switching capabilities.
  Part 2: In this part, the child alternates between numbers and letters (e.g., 1-A-2-B), which adds a layer of complexity to assess cognitive flexibility and visual-motor coordination.
Forward Digit Span | 8 weeks
  Measures the ability to temporarily hold and recall sequences of numbers in the same order they are presented, assessing short-term memory
Backward Digit Span | 8 weeks
  Requires the child to recall sequences of numbers in reverse order, testing their working memory and cognitive processing capabilities.
Digit Sequencing | 8 weeks
  Involves recalling a series of digits in numerical order, further assessing the ability to manipulate and reorganize information in working memory
Inhibitory Control and Cognitive Flexibility | 8 weeks
  tested by Stroop Test This test evaluates the child's ability to inhibit automatic responses and demonstrate cognitive flexibility. In the classic Stroop task, the child must name the ink color of words that are incongruent with their meaning (e.g., the word "red" printed in blue ink). It measures how well the child can control their impulsive responses and manage conflicting information.

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Ahmed Awan Principal Investigator, phD, Principal Investigator — Riphah International University
Locations (1):
- Different Schools, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No